CLINICAL TRIAL: NCT00741143
Title: Effect of Iron Fortified Wheat Flour on Cognition and Iron Status in Indian School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. John's Research Institute (Other)
Collaborators: Akzo Nobel (Industry); Ministry of Science and Technology, India (Other Government)
Responsible Party: Dr Sumithra Muthayya, St Johns Research Institute
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: SJRI-BT-PR-8947; BT/PR-8947/FNS/20/325/2007
Record Dates: First submitted 2008-08-23; First posted 2008-08-26 (Estimated); Last update posted 2008-08-26 (Estimated); Status verified 2008-08

CONDITIONS: Iron Deficiency; Iron Deficiency Anemia; Cognition
Keywords: Food Fortification; Iron deficiency; NaFeEdta; Iron deficiency anemia; Cognition
MeSH Terms: conditions — Iron Deficiencies; Anemia, Iron-Deficiency | interventions — Fe(III)-EDTA

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Group that receives NaFeEDTA fortified wheat flour
  Interventions: Other: Fortification of wheat flour with NaFeEdta
- 2 (Placebo Comparator): Unfortified wheat flour
  Interventions: Other: Fortification of wheat flour with NaFeEdta

INTERVENTIONS:
Other: Fortification of wheat flour with NaFeEdta — NaFeEdta Fortified Wheat Flour (100g)provided as a lunch meal. Fortification level of 6mg Fe/100g/day/child for 7 months

SUMMARY:
This study is designed to evaluate the efficacy of NaFeEDTA-fortified whole wheat flour in improving cognition, hemoglobin, iron status and total body iron among school children in urban Bangalore.

DETAILED DESCRIPTION:
Background: Iron (Fe) deficiency is a major cause of anemia in children. Fortification of wheat flour with NaFeEDTA, a highly bioavailable iron fortificant that protects Fe from the phytic acid present in wheat flour, could be a practical approach to addressing this problem.

Aims: To evaluate the efficacy of NaFeEDTA-fortified whole wheat flour in improving mental performance and reducing iron deficiency and improving body iron stores in urban, school going Indian children.

Methods: A randomized, double-blind, 7 month, school-based feeding trial was carried out in Bangalore, India. Iron-depleted (serum ferritin, SF <20 µg/L), and/or iron deficient (serum transferrin receptor, TfR >7.6 mg/L), 6 -13 year old children (N=194) were randomly assigned to either receive a whole wheat flour based lunch meal fortified with 6 mg Fe as NaFeEDTA or an identical unfortified control meal. The meals were administered under supervision and left overs were weighed. Hemoglobin (Hb) and iron status were measured at baseline, 3.5 months, and 7 months. At baseline and at 7 months, the study children were also subjected to a battery of cognitive tests to assess attention/concentration, motor development, visuospatial and verbal abilities. Sensory evaluation using triangle tests were carried out using meals prepared from the fortified and unfortified whole wheat flour.

ELIGIBILITY:
Inclusion Criteria:

* Children with depleted iron stores (serum ferritin < 20 µg/L or iron deficiency serum transferrin receptor >7.6 mg/L)

Exclusion Criteria:

* Hb < 8g/dl, any metabolic illness, use of medication, on iron supplementation

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 194 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
change in cognitive abilities | 7 months

SECONDARY OUTCOMES:
changes in iron status indicators | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Sumithra Muthayya, PhD, Principal Investigator — St Johns Research Institute, Sarjapur Road, Bangalore
Locations (1):
- St Johns Research Institute, Bangalore, Karnataka, India

REFERENCES:
- [Derived] Muthayya S, Thankachan P, Hirve S, Amalrajan V, Thomas T, Lubree H, Agarwal D, Srinivasan K, Hurrell RF, Yajnik CS, Kurpad AV. Iron fortification of whole wheat flour reduces iron deficiency and iron deficiency anemia and increases body iron stores in Indian school-aged children. J Nutr. 2012 Nov;142(11):1997-2003. doi: 10.3945/jn.111.155135. Epub 2012 Sep 26. PMID 23014487